CLINICAL TRIAL: NCT02318719
Title: An Asian, Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled 14-Week Study of DS-5565 in Patients With Post-herpetic Neuralgia Followed by a 52-Week Open-label Extension
Brief Title: DS-5565 Phase III Study for Post-herpetic Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: SRL Medisearch Inc. (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS5565-A-J304
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Post-Herpetic Neuralgia
Keywords: Post-Herpetic Neuralgia; Developmental Phase III
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — mirogabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (14-weeks)
  Interventions: Drug: Placebo
- DS-5565 15 mg Group (Experimental): DS-5565 15 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Interventions: Drug: DS-5565
- DS-5565 20 mg Group (Experimental): DS-5565 20 mg, oral administration, Treatment period; 1-week titration and 13-weeks fixed dose
  Interventions: Drug: DS-5565
- DS-5565 30 mg Group (Experimental): DS-5565 30 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Interventions: Drug: DS-5565

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: DS-5565
  Other Names: Mirogabalin
  Arms: DS-5565 15 mg Group; DS-5565 20 mg Group; DS-5565 30 mg Group

SUMMARY:
Investigate the efficacy and safety of DS-5565 in subjects with Post-Herpetic Neuralgia (PHN) in comparison to placebo

DETAILED DESCRIPTION:
[Double Blind Phase] The primary objective is to compare change in the Average Daily Pain Score (ADPS) from baseline to Week 14 in Asian subjects with PHN receiving DS-5565 versus placebo.

[Open Extension Phase] The objective is to assess the long-term safety and efficacy of DS-5565 in subjects with PHN.

ELIGIBILITY:
Inclusion Criteria:

* PHN defined as pain present for more than 3 months after herpes zoster skin rash at screening
* At screening, a pain scale of ≥ 40 mm

Exclusion Criteria:

* Previous use of neurolytic block

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daichii Sankyo
Locations (1):
- Medical Corporation Fujigaki Clinic, Ōita, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Kato J, Baba M, Kuroha M, Kakehi Y, Murayama E, Wasaki Y, Ohwada S. Safety and Efficacy of Mirogabalin for Peripheral Neuropathic Pain: Pooled Analysis of Two Pivotal Phase III Studies. Clin Ther. 2021 May;43(5):822-835.e16. doi: 10.1016/j.clinthera.2021.03.015. Epub 2021 May 29. PMID 34059327
- [Derived] Kato J, Matsui N, Kakehi Y, Murayama E, Ohwada S. Long-term safety and efficacy of mirogabalin in Asian patients with postherpetic neuralgia: Results from an open-label extension of a multicenter randomized, double-blind, placebo-controlled trial. Medicine (Baltimore). 2020 Sep 4;99(36):e21976. doi: 10.1097/MD.0000000000021976. PMID 32899037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 765 participants who met all inclusion and no exclusion criteria were enrolled in the study; 763 participants received treatment in the double-blind phase. A total of 239 participants received treatment in the open-label extension phase.
Pre-assignment Details: This study included a double-blind phase where participants received DS-5565 (15 mg, 20 mg, or 30 mg) or placebo and an open-label extension phase where participants received DS-5565 (starting dose 5 mg).
Groups:
- Placebo: Participants who received placebo for 14 weeks.
- DS-5565 15 mg/Day: Participants received oral administrations of DS-5565 15 mg/day with a 2 week titration (5 mg/day during 1st week and 10 mg/day during 2nd week) followed by 12 weeks fixed dose (15 mg/day).
- DS-5565 20 mg/Day: Participants received oral administrations of DS-5565 20 mg/day with a 1 week titration (5 mg BID) followed by 13 weeks fixed dose (10 mg BID).
- DS-5565 30 mg/Day: Participants received oral administrations of DS-5565 30 mg/day with a 2 week titration (5 mg BID during 1st week and 10 mg BID during 2nd week) followed by 12 weeks fixed dose (15 mg BID).
- DS-5565 Open-label Extension: Participants who received 5 mg BID for the first 2 weeks and 10 mg BID for the second 2 weeks (i.e., Week 3 and 4). At Week 5, the dosage escalated to 15 mg BID if there were no concerns in safety. For the subsequent visits, the dosage may have changed to either 10 mg BID or 15 mg BID depending on safety findings.
Period: Double-blind Phase
Arm/Group | Placebo | DS-5565 15 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day | DS-5565 Open-label Extension
Started | 304 | 153 | 153 | 155 | 0
Did Not Receive Treatment | 1 | 1 | 0 | 0 | 0
Completed | 266 | 137 | 128 | 140 | 0
Not Completed | 38 | 16 | 25 | 15 | 0
Not completed — Adverse Event | 7 | 6 | 12 | 4 | 0
Not completed — Lack of Efficacy | 5 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 7 | 9 | 10 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0
Period: Open-label Extension Phase
Arm/Group | Placebo | DS-5565 15 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day | DS-5565 Open-label Extension
Started | 0 | 0 | 0 | 0 | 239 (A portion of participants who completed the double-blind phase enrolled in the open-label extension.)
Completed | 0 | 0 | 0 | 0 | 184
Not Completed | 0 | 0 | 0 | 0 | 55
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 15
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 31
Not completed — Other | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- DS-5565 15 mg: Participants who received oral administration of DS-5565 15 mg with a 2 week titration and 12 weeks fixed dose treatment period.
- DS-5565 20 mg: Participants who received oral administration of DS-5565 20 mg with a 1 week titration and 13 weeks fixed dose treatment period.
- DS-5565 30 mg: Participants who received oral administration of DS-5565 30 mg with a 2 week titration and 12 weeks fixed dose treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | DS-5565 15 mg | DS-5565 20 mg | DS-5565 30 mg | Total
Number analyzed (Participants) | 304 | 153 | 153 | 155 | 765
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 47 | 39 | 64 | 252
  >=65 years | 202 | 106 | 114 | 91 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.13) | 66.6 (8.97) | 68.9 (9.19) | 64.5 (10.74) | 66.5 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 56 | 62 | 59 | 304
  Male | 177 | 97 | 91 | 96 | 461
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 304 | 153 | 153 | 155 | 765
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 304 | 153 | 153 | 155 | 765

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average Daily Pain Score (ADPS) From Baseline to Week 14 Following Oral Administration of DS-5565 in Asian Participants With Post-herpetic Neuralgia
Description: Each participant recorded a pain score in the electronic patient diary once daily from the day after the screening visit (Visit 1) to the end of treatment/early termination visit (Visit 10). Prior to taking the study drug each morning, the participant selected the number that best described his or her pain over the past 24 hours on a scale of 0 (no pain) to 10 (worst possible pain). Higher ADPS scores indicated worse outcome. ADPS was the weekly average pain score based on the pain scores from the electronic patient diaries (Pain diary).
  In this outcome, the change from baseline in ADPS is being reported with negative values representing improvements in average daily pain. The larger the negative value (ie. improvement), the greater the improvement in average daily pain.
Time Frame: Baseline to Week 14
Population: Average daily pain score (ADPS) was assessed in the modified Intent-to-Treat Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | DS-5565 15 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day
Number analyzed (Participants) | 303 | 152 | 153 | 155
units on a scale
  Week 1 | -0.10 (0.743) | -0.39 (0.787) | -0.54 (0.783) | -0.46 (0.693)
  Week 2 | -0.33 (0.902) | -0.72 (1.036) | -1.06 (0.998) | -0.95 (1.003)
  Week 3 | -0.48 (1.030) | -0.96 (1.195) | -1.16 (1.122) | -1.20 (1.188)
  Week 4 | -0.64 (1.163) | -1.08 (1.283) | -1.24 (1.192) | -1.33 (1.236)
  Week 5 | -0.74 (1.215) | -1.17 (1.351) | -1.36 (1.233) | -1.49 (1.275)
  Week 6 | -0.81 (1.329) | -1.29 (1.412) | -1.44 (1.337) | -1.55 (1.277)
  Week 7 | -0.96 (1.399) | -1.32 (1.409) | -1.45 (1.382) | -1.67 (1.346)
  Week 8 | -1.03 (1.466) | -1.39 (1.509) | -1.40 (1.455) | -1.62 (1.375)
  Week 9 | -1.09 (1.478) | -1.44 (1.574) | -1.42 (1.480) | -1.72 (1.431)
  Week 10 | -1.15 (1.547) | -1.49 (1.632) | -1.51 (1.564) | -1.81 (1.486)
  Week 11 | -1.22 (1.601) | -1.53 (1.647) | -1.60 (1.576) | -1.84 (1.473)
  Week 12 | -1.21 (1.614) | -1.59 (1.727) | -1.63 (1.624) | -1.89 (1.519)
  Week 13 | -1.25 (1.665) | -1.63 (1.769) | -1.68 (1.643) | -1.95 (1.486)
  Week 14 | -1.31 (1.710) | -1.67 (1.717) | -1.73 (1.715) | -1.96 (1.501)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg/Day; Placebo vs DS-5565 15 mg/day at Week 14; Test type: Superiority; p = 0.0170, Mixed Models Analysis — DS-5565 20 mg and 30 mg vs placebo were tested at level of 0.025. If both were significant, 15 mg was tested at 0.05. If neither were significant, 15 mg was no longer tested. If either 20 mg or 30 mg was significant, 15 mg was tested at 0.025; Difference of least square mean = -0.41, 95% CI 2-sided [-0.74 to -0.07]
Statistical Analysis 2: Comparison: Placebo vs DS-5565 20 mg/Day; Placebo vs DS-5565 20 mg/day at Week 14; Test type: Superiority; p = 0.0058, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of least square means = -0.47, 95% CI 2-sided [-0.81 to -0.14]
Statistical Analysis 3: Comparison: Placebo vs DS-5565 30 mg/Day; Placebo vs DS-5565 30 mg/day at Week 14; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of least square means = -0.77, 95% CI 2-sided [-1.10 to -0.44]

2. Secondary Outcome: Change in Visual Analog Scale (VAS) Pain From Baseline (Week 14) to Week 66 Following Administration of DS-5565 in Asian Participants With Post-herpetic Neuralgia
Description: Visual Analog Scale (VAS) pain is a 10-point assessment tool to measure pain levels, where 0 is defined as 'no pain' and 10 is defined as 'worst possible pain'. Higher VAS pain scores indicate worse outcome.
  In this outcome, the change from baseline in VAS pain is being reported with negative values representing improvements in pain intensity. The larger the negative value (ie. improvement), the greater the improvement in pain intensity.
Time Frame: From baseline (Week 14) to Week 66
Population: Visual analog scale (VAS) was assessed in the modified Intent-to-Treat Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DS-5565 Open-label Extension
Number analyzed (Participants) | 237
units on a scale
  Week 16 | -0.70 (9.530)
  Week 18 | 4.60 (9.850)
  Week 22 | -8.30 (12.070)
  Week 26 | -8.60 (12.030)
  Week 30 | -8.70 (13.670)
  Week 34 | -10.00 (14.260)
  Week 38 | -10.40 (14.450)
  Week 42 | -11.20 (13.930)
  Week 46 | -12.00 (13.890)
  Week 50 | -12.60 (14.530)
  Week 54 | -12.50 (14.760)
  Week 58 | -12.90 (15.250)
  Week 62 | -14.00 (16.790)
  Week 66 | -14.70 (15.270)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from after the participant signed the informed consent form and up to 7 days after the last dose of the study drug (the post-treatment follow-up visit [Visit 11]), up to 2 years 5 months.
Description: Treatment-emergent AEs were defined as any AEs that appeared after the first administration of study treatment or that worsened relative to the pre-treatment state. Safety data were reported from participants in the Safety Analysis Set who had available safety data; 2 participants in the DS-5565 open-label extension data did not have available safety data and were not included in the analysis.
Arm/Group | Placebo | DS-5565 15 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day | DS-5565 Open-label Extension
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/152 | 0/153 | 0/155 | 1/237
Serious Adverse Events (participants affected / at risk) | 0/303 | 0/152 | 0/153 | 0/155 | 20/237
Other Adverse Events (participants affected / at risk) | 45/303 | 44/152 | 53/153 | 72/155 | 99/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=303) | DS-5565 15 mg/Day (N=152) | DS-5565 20 mg/Day (N=153) | DS-5565 30 mg/Day (N=155) | DS-5565 Open-label Extension (N=237)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dissociative disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Uterine fibrosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Large intestinal polypectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Nasal polypectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=303) | DS-5565 15 mg/Day (N=152) | DS-5565 20 mg/Day (N=153) | DS-5565 30 mg/Day (N=155) | DS-5565 Open-label Extension (N=237)
Nasopharyngitis (Infections and infestations) | 26 | 13 | 16 | 20 | 39
Somnolence (Nervous system disorders) | 11 | 20 | 26 | 37 | 36
Dizziness (Nervous system disorders) | 10 | 10 | 15 | 24 | 26
Oedema (General disorders) | 2 | 2 | 6 | 11 | 14
Weight increased (Investigations) | 1 | 7 | 8 | 8 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT02318719/Prot_SAP_000.pdf